CLINICAL TRIAL: NCT01271010
Title: Prospective Study of Efficacy and Safety of RFC (Rituximab, Fludarabine, Cyclophosphamide) Regimen as a First-Line Therapy in Patients With B-Cell Chronic Lymphocytic Leukemia and Favorable Somatic Status
Brief Title: A Study of Rituximab in Combination With Fludarabine and Cyclophosphamide in Participants With Chronic Lymphocytic Leukemia and Favorable Somatic Status
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25136
Record Dates: First submitted 2011-01-04; First posted 2011-01-06 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2017-08

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; fludarabine; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rituximab + Fludarabine + Cyclophosphamide (Experimental): Participants received rituximab 375 milligrams per square meter (mg/m^2) intravenously (IV) on Day 1 of Cycle 1, then 500 mg/m^2 IV on Day 1 of each subsequent cycle; fludarabine 25 mg/m^2 IV or 40 mg/m^2 orally on Days 1-3 of each cycle and cyclophosphamide 250 mg/m^2 IV or 250 mg/m^2 orally on Days 1-3 of each cycle. Treatment duration was 6 cycles, 28 days each.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Rituximab

INTERVENTIONS:
Drug: Cyclophosphamide — Participants received cyclophosphamide 250 mg/m^2 IV or 250 mg/m^2 orally on Days 1-3 of each cycle.
Drug: Fludarabine — Participants received fludarabine 25 mg/m^2 IV or 40 mg/m^2 orally on Days 1-3 of each cycle.
Drug: Rituximab — Participants received 375 mg/m^2 IV on Day 1 of Cycle 1, then 500 mg/m^2 IV on Day 1 of each subsequent cycle.
  Other Names: MabThera

SUMMARY:
This multi-center, single-arm study evaluated the efficacy and safety of rituximab in combination with fludarabine and cyclophosphamide in participants with B-cell chronic lymphocytic leukemia (CLL) and favorable somatic status.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of previously untreated B-cell CLL confirmed immunophenotypically
* For participants, age 60-70 years: Cumulative Illness Rating Scale (CIRS) comorbidity score less than or equal to (</=) 6
* Binet stage B, C or A with progression
* Life expectancy greater than or equal to (>/=) 12 months
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Women of child bearing potential and men should agree to use highly reliable contraceptive method throughout the treatment period and within 12 months after treatment completion

Exclusion Criteria:

* Participants with small-cell lymphoma
* Participants with auto-immune hemolytic anemia
* Concomitant malignant disease during enrollment, except basal cell carcinoma of the skin
* Chemotherapy for concomitant malignant disease given within 12 months prior to study enrollment
* Participants with Richter's Syndrome
* Participants with symptomatic Hepatitis B infection
* Any clinically significant infection that could not be cured prior to enrollment, including Human Immunodeficiency Virus (HIV) infection
* Creatinine clearance less than (<) 30 milliliters per minute (mL/min)
* Participants with congestive heart failure (CHF) New York Heart Association (NYHA) III-IV
* Participants with liver failure and acute hepatitis of any etiology
* Any other medical or mental condition which may preclude from receiving the entire course of protocol specified treatment or signing the informed consent
* History of an anaphylactic reaction to murine antibodies, proteins, or any other ingredient of rituximab
* Pregnancy and breast-feeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2011-06-17 (Actual); Primary Completion 2016-05-04 (Actual); Study Completion 2016-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Russia (10):
  - The order of Honour pin Irkutsk regional clinical hospital; Hematology Department, Irkutsk
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - Regional Clinical Oncology Despensary #1; Hematology Department, Krasnodar
  - N.N.Blokhin Russian Cancer Research Center; Dept. of Chemotherapy & Hemoblastosis, Moscow
  - City Clinical Hospital After Botkin; Hematology, Moscow
  - Saint-Petersburg SHI City Clinical Hospital #31, Saint Petersburg
  - City Clinical Hospital #15; Hematology department, Saint Petersburg
  - Leningrad Regional Clinical Hospital; Hematology #1, Saint Petersburg
  - GUZ Tula Regioanal Clinical Hospital; Hematology, Tula
  - Republican clinical hospital named after G.G. Kuvatov, Ufa

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Started | 89
Completed | 28
Not Completed | 61
Not completed — Reason not specified | 11
Not completed — Start of new CLL therapy | 1
Not completed — Protocol Violation | 1
Not completed — Death | 2
Not completed — Progression and relapse of disease | 1
Not completed — Withdrawal by Subject | 18
Not completed — Disease progression | 27

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (6.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 58

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Remission
Description: Complete remission was defined as the disappearance of all signs of disease.
Time Frame: Up to approximately 5 years
Population: All enrolled participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 73
percentage of participants | 49.3

2. Primary Outcome: Percentage of Participants With Disease Progression
Description: Disease progression was defined as an increase in lymphocytosis, or enlargement of the lymph nodes or spleen.
Time Frame: Up to approximately 5 years
Population: All enrolled participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 73
percentage of participants | 5.5

3. Primary Outcome: Percentage of Participants With Stable Disease
Description: Stable disease was defined as not meeting the criteria for partial remission or disease progression
Time Frame: Up to approximately 5 years
Population: All enrolled participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 73
percentage of participants | 4.1

4. Primary Outcome: Percentage of Participants With Partial Remission
Description: Partial remission was defined as a reduction in tumor size by >50%.
Time Frame: Up to approximately 5 years
Population: All enrolled participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 73
percentage of participants | 41.1

5. Primary Outcome: Duration of Response
Description: Duration of Response was defined as the time period from the last day of study treatment to the day when disease progression occurred in participants who previously had complete or partial remission. Disease progression was defined as an increase in lymphocytosis, or enlargement of the lymph nodes or spleen. Complete remission was defined as the disappearance of all signs of disease. Partial remission was defined as a reduction in tumor size by >50%.
Time Frame: Up to approximately 5 years
Population: Enrolled participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 61
days | NA [NA to NA] — Median of duration of response to treatment was not achieved.

6. Primary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time period from the first day of study treatment to the day when disease progression occurred. Disease progression was defined as an increase in lymphocytosis, or enlargement of the lymph nodes or spleen.
Time Frame: Up to approximately 5 years
Population: Enrolled participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 85
days | NA [NA to NA] — Median of progression-free survival was not achieved.

7. Primary Outcome: Event-free Survival
Description: Event-free survival was defined as the time period from the first day of study treatment to occurrence of any of the following events: appearance of disease progression or relapse; prescription of a new treatment for disease relapse; death caused by B-cell chronic lymphocytic leukemia (B-CLL); or complications from B-CLL or therapy. Relapse was defined as disease progression in participants with complete or partial remission lasting at least 6 months after treatment completion. Disease progression was defined as an increase in lymphocytosis, or enlargement of the lymph nodes or spleen. Complete remission was defined as the disappearance of all signs of disease. Partial remission was defined as a reduction in tumor size by >50%.
Time Frame: Up to approximately 5 years
Population: Enrolled participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 85
days | 1567 [1036 to NA] — The curve representing the upper confidence limit for the survivor function was above 0.75. Therefore, the upper confidence limit could not be estimated.

8. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time period from the first day of study treatment to participant death.
Time Frame: Up to approximately 5 years
Population: Enrolled participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 89
days | NA [NA to NA] — Median and confidence intervals were not calculable due to the low number of events of death.

9. Primary Outcome: Percentage of Participants With Phenotypic Remission
Description: Phenotypic remission was considered achieved if a participant had a negative test for minimal residual disease. A negative test for minimal residual disease was defined as tumor cells ≤0.01% of the total number of peripheral leukocytes.
Time Frame: Up to approximately 5 years
Population: Enrolled participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 63
percentage of participants | 66.7

10. Primary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious AEs
Description: An AE was defined as any unfavorable medical occurrence in a participant receiving a study drug, regardless of relationship the study drug. An AE was considered serious if it met any of the following criteria: was fatal or life-threatening; required hospitalization or prolonged hospitalization; led to persistent or significant disability/incapacity; was a congenital anomaly/birth defect; was clinically significant and/or required an intervention to prevent any of the listed criteria.
Time Frame: Up to approximately 5 years
Population: All enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 89
percentage of participants
  Non-serious AEs | 78.65
  Serious AEs | 13.48

ADVERSE EVENTS:
Time Frame: Up to approximately 5 years
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 12/89
Other Adverse Events (participants affected / at risk) | 70/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Fludarabine + Cyclophosphamide (N=89)
Herpes zoster (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Proctitis infectious (Infections and infestations) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Squamous cell carcinoma of lung (Respiratory, thoracic and mediastinal disorders) | 1
Agranulocytosis (Blood and lymphatic system disorders) | 1
Neuroendocrine tumour (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Brain contusion (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Contusion (Musculoskeletal and connective tissue disorders) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Duodenal ulcer haemorrhage (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Fludarabine + Cyclophosphamide (N=89)
Neutrophil count decreased (Investigations) | 37
White blood cell count decreased (Investigations) | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Anaemia (Blood and lymphatic system disorders) | 9
Leukocytosis (Blood and lymphatic system disorders) | 5
Respiratory tract infection (Infections and infestations) | 8
Nausea (Gastrointestinal disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.